CLINICAL TRIAL: NCT01468896
Title: A Phase I/II Trial of Cetuximab in Combination With Interleukin-12 Administered to Patients With Unresectable Primary or Recurrent Squamous Cell Carcinoma of the Head and Neck
Brief Title: Cetuximab and Recombinant Interleukin-12 in Treating Patients With Squamous Cell Carcinoma of the Head and Neck That is Recurrent, Metastatic, or Cannot Be Removed by Surgery
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-03631; NCI-2011-03631 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2011C0019; 11010; CDR0000715306; 8860 (Other: Ohio State University Comprehensive Cancer Center); 8860 (Other: CTEP); N01CM00070 (NIH); P30CA016058 (NIH); U01CA076576 (NIH); UM1CA186712 (NIH)
Record Dates: First submitted 2011-11-08; First posted 2011-11-10 (Estimated); Results first posted 2017-08-31 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Head and Neck Squamous Cell Carcinoma; Recurrent Head and Neck Squamous Cell Carcinoma; Unresectable Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab; (225)Ac-DOTA-c(RGDyK); Interleukin-12; Interleukin-12 Subunit p35

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (cetuximab and recombinant interleukin-12) (Experimental): Patients receive cetuximab IV over 1-2 hours on day 1 and recombinant interleukin-12 SC on days 2 and 5 beginning in course 2. Treatment repeats every 2 weeks for 12 courses in the absence of disease progression or unacceptable toxicity. Patients achieving clinical response or stable disease may continue with therapy until disease progression.
  Interventions: Biological: Cetuximab; Biological: Edodekin alfa; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Cetuximab — Given IV
  Other Names: C 225; C-225; C225; Cetuximab Biosimilar CDP-1; Cetuximab Biosimilar CMAB009; Cetuximab Biosimilar KL 140; Chimeric Anti-EGFR Monoclonal Antibody; Chimeric MoAb C225; Chimeric Monoclonal Antibody C225; Erbitux; IMC-C225
Biological: Edodekin alfa — Given SC
  Other Names: Cytotoxic Lymphocyte Maturation Factor; IL-12; Interleukin 12; Interleukin-12; Natural Killer Cell Stimulatory Factor; NM-IL-12; Recombinant human interleukin-12 (IL-12) cytokine; Ro 24-7472
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I/II trial studies the side effects and best dose of recombinant interleukin-12 when given together with cetuximab and to see how well they work in treating patients with squamous cell carcinoma of the head and neck that has come back, spread to another place in the body, or cannot be removed by surgery. Recombinant interleukin-12 may stimulate the white blood cells to kill tumor cells. Immunotherapy with monoclonal antibodies, such as cetuximab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread Giving recombinant interleukin-12 together with cetuximab may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To find a safe and tolerable interleukin (IL)-12 (recombinant interleukin-12) dose for use in combination with cetuximab in patients with squamous cell carcinoma of the head and neck. (Phase I) II. To determine the response rate to the combination of IL-12 and cetuximab. (Phase II)

SECONDARY OBJECTIVES:

I. To characterize the immunologic effects of IL-12 when administered in combination with cetuximab.

OUTLINE: This is a phase I, dose-escalation study of recombinant IL-12 followed by a phase II study.

Patients receive cetuximab intravenously (IV) over 1-2 hours on day 1 and recombinant interleukin-12 subcutaneously (SC) on days 2 and 5 beginning in course 2. Treatment repeats every 2 weeks for 12 courses in the absence of disease progression or unacceptable toxicity. Patients achieving clinical response or stable disease may continue with therapy until disease progression.

After completion of study treatment, patients are followed up for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically-proven recurrent and/or metastatic squamous cell carcinoma of the head and neck that is unresectable; patients in the phase II portion of the trial must have measurable disease
* Any number of prior systemic therapies for metastatic/recurrent disease are permitted in both the phase I and II portions of the study; patients need not have received a prior cetuximab-based chemotherapy regimen to be eligible for this trial
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 6 months
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 times upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* The effects of IL-12 on the developing human fetus are unknown; for this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents
* Patients with known brain metastases may be enrolled if this site of disease has been adequately treated, the patient does not require steroids, and the patient has been stable for at least 3 months prior to enrollment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to IL-12 or other agents used in study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because IL-12 is an agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with IL-12, breastfeeding should be discontinued if the mother is treated with IL-12; these potential risks may also apply to other agents used in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-10-26 (Actual); Primary Completion 2015-09-29 (Actual); Study Completion 2026-03-19 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: William E Carson, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (2):
- United States (2):
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 (Phase I): Cetuximab 500 mg/m2 i.v. on day 1 of the two week cycle followed by subcutaneous IL-12 (Dose Escalation) on days 2 and 5 of the 2 week cycle, beginning with cycle 2.
- Arm II (Phase II): Cetuximab 500 mg/m2 i.v. on day 1 of the two week cycle followed by subcutaneous IL-12 at the MTD on days 2 and 5 of the 2 week cycle beginning with cycle 2. No IL-12 is given in the first cycle. IL-12 dosing will begin in cycle 2. The IL-12 dose is 0.3 mcg/kg.
Period: Overall Study
Arm/Group | Arm 1 (Phase I) | Arm II (Phase II)
Started | 6 | 17
Completed | 6 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 1 (Phase 1): Cetuximab 500 mg/m2 i.v. on day 1 of the two week cycle followed by subcutaneous IL-12 (Dose Escalation) on days 2 and 5 of the 2 week cycle, beginning with cycle 2.
- Total: Total of all reporting groups
Arm/Group | Arm 1 (Phase 1) | Arm II (Phase II) | Total
Number analyzed (Participants) | 6 | 17 | 23
Age, Continuous [Median (Full Range); unit: years] | 56.5 [52 to 64] | 62 [51 to 84] | 61 [51 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 5 | 17 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 16 | 22
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 5 | 14 | 19
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 17 | 23

OUTCOME MEASURES:

1. Primary Outcome: Number of Dose-limiting Toxicity Incidents to Determine the Maximum Tolerated Dose of IL-12, Evaluated Using the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0 (Phase I)
Time Frame: 14 days
Measure: Number; unit: Dose limiting toxicities
Arm/Group | Arm 1 (Phase I) | Arm II (Phase II)
Number analyzed (Participants) | 6 | 17
Dose limiting toxicities | 2 | 0

2. Primary Outcome: Proportion of Patients Who Have Any Response to Treatment (Complete Response or Partial Response), Determined According to Response Evaluation Criteria in Solid Tumors (Phase II)
Description: The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Ninety percent confidence intervals for the true success proportion will be calculated according to the approach of Duffy and Santner. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 6 months
Measure: Number; unit: proportion of patients
Arm/Group | Arm II (Phase II)
Number analyzed (Participants) | 17
proportion of patients | 0

3. Secondary Outcome: Induction of Systemic Plasma Levels of Interferon-gamma
Description: Explores graphically how changes in this marker differ between those with versus without an objective response to therapy as well as other potential factors.
Time Frame: Baseline up to day 50
Population: Unable to compare the plasma levels of interferon-gamma between those with versus without an objective response to therapy due to no objective response seen for Phase I or Phase II patients.
Arm/Group | Arm 1 (Phase I) | Arm II (Phase II)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Confirmed Clinical Responses (Phase I)
Description: Summarized by simple descriptive summary statistics. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 (Phase I)
Number analyzed (Participants) | 6
Participants | 0

5. Secondary Outcome: Overall Survival (Phase II)
Description: The Kaplan-Meier method will be used to estimate overall survival distribution.
Time Frame: From the date of registration to date of death, assessed up to 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1 (Phase I) | Arm II (Phase II)
Number analyzed (Participants) | 0 | 17
months |  | 10.6 [5.3 to 12.7]

6. Secondary Outcome: Proportion of Patients Who Are Progression-free (Phase I)
Description: as for outcome 4
Time Frame: 6 months
Measure: Number; unit: proportion of patients
Arm/Group | Arm 1 (Phase I) | Arm II (Phase II)
Number analyzed (Participants) | 6 | 0
proportion of patients | .17 |

7. Secondary Outcome: Time to Disease Progression (Phase II)
Description: The Kaplan-Meier method will be used to estimate time to progression distributions.
Time Frame: From date of registration to date of progression, assessed up to 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1 (Phase I) | Arm II (Phase II)
Number analyzed (Participants) | 0 | 17
months |  | 4.6 [1.8 to 13.3]

ADVERSE EVENTS:
Description: Toxicities were graded using the National Cancer Institutes Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Arm/Group | Arm 1 (Phase I) | Arm II (Phase II)
Serious Adverse Events (participants affected / at risk) | 5/6 | 9/17
Other Adverse Events (participants affected / at risk) | 6/6 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (Phase I) (N=6) | Arm II (Phase II) (N=17)
General Disorders and administration site conditions (General disorders) | 1 (1) | 0 (0)
Arterial Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Neoplasm benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — includes cysts and polyps
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (Phase I) (N=6) | Arm II (Phase II) (N=17)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (7) | 6 (7)
Skin and subcutaneous tissue disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5) — other
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (3) | 6 (28)
Hyponatremia (Metabolism and nutrition disorders) | 2 (3) | 5 (15)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (4) | 5 (17)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3) | 2 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 9 (17)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (4) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 3 (5)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Fatigue (General disorders) | 4 (4) | 8 (13)
Chills (General disorders) | 0 (0) | 5 (5)
Fever (General disorders) | 1 (1) | 4 (8)
Edema Face (General disorders) | 0 (0) | 2 (2)
Edema Limbs (General disorders) | 1 (1) | 1 (1)
Flu Like Symptoms (General disorders) | 0 (0) | 2 (2)
Malaise (General disorders) | 0 (0) | 2 (2)
General disorders and administration site conditions-other (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (9) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (3)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatuelence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal Disorder-other (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomach Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (4)
Lymphocyte count decreased (Investigations) | 6 (10) | 6 (18)
Alanine aminotransferase increased (Investigations) | 4 (6) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 3 (5) | 5 (11)
Alkaline phosphatase increased (Investigations) | 2 (3) | 3 (9)
White blood cell decreased (Investigations) | 1 (1) | 4 (18)
Weight loss (Investigations) | 0 (0) | 4 (8)
Weight gain (Investigations) | 0 (0) | 2 (10)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (4)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 5 (6)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3)
Facial muscle weakness (Nervous system disorders) | 0 (0) | 1 (1)
Facial nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 10 (10) — including cysts and polyps
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonthorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 6 (8)
Hypertension (Vascular disorders) | 1 (1) | 6 (21)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 2 (2)
Skin Infection (Infections and infestations) | 0 (0) | 2 (2)
Esophageal infection (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective disorder-other (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Arterial injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intestinal stoma site bleeding (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Renal and urinary disorders-other (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less